CLINICAL TRIAL: NCT04294966
Title: Age-Related Effects of THC
Acronym: ART
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: University of Chicago (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: IRB20-0112
Record Dates: First submitted 2020-02-27; First posted 2020-03-04 (Actual); Results first posted 2023-11-09 (Actual); Last update posted 2023-11-09 (Actual); Status verified 2023-11

CONDITIONS: Tolerance; Adolescent Behavior; THC
MeSH Terms: conditions — Adolescent Behavior | interventions — Glucose; Dronabinol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (3):
- Placebo (Placebo Comparator)
  Interventions: Drug: Dextrose
- 7.5 mg THC (Active Comparator)
  Interventions: Drug: Dronabinol
- 15 mg THC (Active Comparator)
  Interventions: Drug: Dronabinol

INTERVENTIONS:
Drug: Dextrose — Administering dextrose to healthy volunteers for our placebo group
  Arms: Placebo
Drug: Dronabinol — THC (Marinol® [dronabinol]; Solvay Pharmaceuticals) will be orally administered in doses of 7.5 mg and 15 mg, in opaque capsules with dextrose filler. Placebo capsules contain only dextrose. These doses of THC are known to produce performance impairments as well as subjective intoxication with little to no adverse reactions in experienced occasional, but non-daily cannabis users.
  Arms: 7.5 mg THC
Drug: Dronabinol — THC (Marinol® [dronabinol]; Solvay Pharmaceuticals) will be orally administered in doses of 7.5 mg and 15 mg, in opaque capsules with dextrose filler. Placebo capsules contain only dextrose. These doses of THC are known to produce performance impairments as well as subjective intoxication with little to no adverse reactions in experienced occasional, but non-daily cannabis users.
  Arms: 15 mg THC

SUMMARY:
Increased accessibility to cannabis and its primary psychoactive constituent THC has raised public health concerns. One major concern surrounds the potential risks associated with acute THC intoxication and who might be most at risk. A second major concern is the need to develop sensitive measures that can detect THC intoxication after recent use and enable robust comparisons of intoxication to determine sources of risk. One potential source of risk is age, specifically during the period of adolescence.

DETAILED DESCRIPTION:
There is limited knowledge on the effects of THC in adolescents vs adults. One recent report compared responses to vaporized cannabis in heavy adolescent vs adult cannabis users and found that the adolescents were less sensitive to the drug on most measures. However, their findings were complicated by several factors: i) the study used vaporized cannabis, which may have other constituents and does not offer full control of the dose, ii) the participants were heavy users, making it difficult to determine the influence of prior drug exposure, and iii) the participants were not drug-free at the time of testing. Prior exposure to THC can lead to tolerance, and adolescents and adults may differ in the rate at which they develop tolerance, consistent with changes in CB1R receptor function. Our study will compare adolescent (here, aged 18 to 20) and adult (here, aged 30 to 40) responses to THC in relatively light cannabis users who are drug-free at the time of testing.

ELIGIBILITY:
Inclusion Criteria:

* 18-20 years old OR 30-40 years old
* Body Mass Index 19-26
* High school education, fluent in English
* Occasional cannabis users ( 0 times in past 30 days AND used cannabis no more than 20 times in lifetime)

Exclusion Criteria:

* History of daily cannabis use
* Past or present severe substance use disorder
* Current or past diagnosis with drug treatment for psychosis/bipolar/schizophrenia
* Cardiovascular illness, high blood pressure, abnormal electrocardiogram
* Current medications
* Pregnant or planning to become pregnant

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2020-03-10 (Actual); Primary Completion 2021-05-01 (Actual); Study Completion 2021-05-01 (Actual)

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - University of Chicago Hospital, Chicago, Illinois
  - University of Chicago, Chicago, Illinois

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Placebo: Dextrose: Administering dextrose to health volunteers for our placebo group
Period: Overall Study
Arm/Group | Placebo | 7.5 mg THC | 15 mg THC
Started | 8 | 8 | 8
Completed | 8 | 8 | 8
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | 7.5 mg THC | 15 mg THC | Total
Number analyzed (Participants) | 8 | 8 | 8 | 24
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 8 | 8 | 8 | 24
  >=65 years | 0 | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 4 | 4 | 12
  Male | 4 | 4 | 4 | 12
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 1 | 1 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 4 | 1 | 1 | 6
  White | 4 | 4 | 4 | 12
  More than one race | 0 | 2 | 2 | 4
  Unknown or Not Reported | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 8 | 8 | 8 | 24

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Profile of Mood States (POMS)
Description: The POMS measures individuals' mood states. This is a validated scale to measure positive and negative mood states. The POMS consists of 72 mood adjectives rated on a Likert scale from 0 (not at all) to 4 (extremely), divided into 8 subscales: Friendliness, Anxiety, Elation, Anger, Fatigue, Depression, Confusion and Vigor, and two composite scales: Positive Mood (Elation minus Depression) and Arousal (Vigor plus Anxiety minus Confusion plus Fatigue). Scoring of this instrument provides a global score of 0 to 120 or individual domain scores of 0 to 20. Lower scores indicate better mood state. The POMS brief form is a simple self-rating instrument.
Time Frame: Through Study Completion, an average of 3 weeks (Baseline - time 0 to Time point 9 (Study Completion))
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | 7.5 mg THC | 15 mg THC
Number analyzed (Participants) | 8 | 8 | 8
units on a scale
  POMS Anxiety Week 1 | 5.75 (5.12) | 12.46 (3.56) | 18.55 (2.55)
  POMS Depression Week 1 | 4.08 (3.60) | 5.05 (3.66) | 6.25 (1.05)
  POMS Vigor Week 1 | 13.00 (6.03) | 8.05 (2.25) | 8.25 (4.25)
  POMS Fatigue Week 1 | 6.67 (6.27) | 14.25 (6.85) | 8.25 (2.55)
  POMS Friendliness Week 1 | 6.42 (3.82) | 16.25 (5.58) | 8.25 (2.22)
  POMS Anxiety Week 3 | 5.50 (4.56) | 14.25 (5.88) | 19.25 (5.22)
  POMS Depression Week 3 | 3.92 (6.64) | 5.28 (1.33) | 8.25 (2.55)
  POMS Vigor Week 3 | 16.83 (5.92) | 6.87 (4.25) | 6.22 (2.22)
  POMS Fatigue Week 3 | 6.0 (4.86) | 8.65 (2.58) | 6.25 (2.55)
  POMS Friendliness Week 3 | 9.42 (5.99) | 8.22 (2.25) | 11.25 (2.25)

ADVERSE EVENTS:
Time Frame: .Through study completion, an average of 3 weeks.
Arm/Group | Placebo | 7.5 mg THC | 15 mg THC
All-Cause Mortality (participants affected / at risk) | 0/8 | 0/8 | 0/8
Serious Adverse Events (participants affected / at risk) | 0/8 | 0/8 | 0/8
Other Adverse Events (participants affected / at risk) | 0/8 | 0/8 | 0/8

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-06-20): https://cdn.clinicaltrials.gov/large-docs/66/NCT04294966/Prot_SAP_000.pdf